CLINICAL TRIAL: NCT01401881
Title: Ischemic Time and Extent of Myocardial Infarction With Cardiac Magnetic Resonance Image in Patients With STEMI and Primary Percutaneous Coronary Intervention Study
Brief Title: Ischemic Time and Extent of Myocardial Infarction (MI) With Cardiac Magnetic Resonance Imaging (CMRI) in Patients With ST Elevation Myocardial Infarction (STEMI) and Primary Percutaneous Coronary Intervention (PCI) Study
Acronym: ITEMMRI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ITEMMRI
Record Dates: First submitted 2010-05-28; First posted 2011-07-25 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post STEMI: The study population will consist of adult patients with acute STEMI and primary PCI with clear identification of symptoms onset, willing to participate in the research protocol and not having any of the exclusion criteria. Patient screening will take place after the primary PCI in the cardiac catheterization laboratory or in the coronary care unit. Participation will be offered to all those who meet eligibility criteria.

SUMMARY:
This study will assess relationship between ischemic time and the extent of myocardial infarction with cardiac magnetic resonance image in patients with STEMI (ST elevation myocardial infarction) and primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background:

Cardiac magnetic resonance image (CMRI) is the preferred method of assessing myocardial infarct size and function. However,the relationship between CMRI changes and the ischemic time [symptom onset to device activation time (S2D)] in patients with primary percutaneous coronary intervention (PCI) is not well understood.

Hypothesis:

The investigators will test the primary hypothesis that there is strong (at least 70%) direct correlation between the S2D time and infarct size by CMRI and inverse correlation with myocardial salvage.

Method:

The investigators will study a prospective cohort of 80 consecutive patients with STEMI and primary PCI. The investigators will perform CMRI at day 3 to 1 post STEMI and a repeat CMRI 30 to 40 days post STEMI.

Exclusion Criteria:

The investigators will exclude patients with 1)-culprit lesion in the distal artery, 2)-glomerular filtration rate (GFR) < 60 mL/min/1.73m2, 3)-pacemaker, defibrillator, aneurysm clips, 4)-body weight > 400lb, 5)-history of allergic reactions to gadlinium based contrast agents, and 6)-those unwilling to participate in the study protocol.

Outcome Measurement:

The primary outcome measure is the CMRI myocardial infarct size (scar). The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.

Follow-up:

Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Clinical features, EKG, cTn elevation, and coronary catheterization findings consistent with an acute STEMI and having primary PCI, with age greater than 18 years, and GFR >= 60 mL/min/1.73m2.

Exclusion Criteria:

1. Renal dysfunction (creatinine clearance < 60 mL/min/1.73m2)
2. Pregnancy or breast-feeding
3. Standard contra-indications to MRI for implanted ferro-magnetic devices - i.e.: pacemakers, defibrillator (AICD), and aneurysm clips
4. Body weight > 400lb
5. Unwilling to participate in the research protocol
6. History of allergic reactions to gadlinium based contrast agents.
7. Too critically ill to receive a MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with acute STEMI and primary PCI with clear identification of symptoms onset, willing to participate in the research protocol and not having any of the exclusion criteria. Patient screening will take place after the primary PCI in the cardiac catheterization laboratory or in the coronary care unit. Participation will be offered to all those who meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
CMRI myocardial infarct size | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The primary outcome measure is the CMRI myocardial infarct size (scar).

SECONDARY OUTCOMES:
CMRI transmurality of scar | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.
CMRI area at risk | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.
CMRI myocardial salvage index | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.
CMRI microvascular obstruction (MVO) | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.
CMRI left ventricle (LV) thrombus | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.
CMRI LV ejection fraction (EF) | Patients will be followed with repeat CMRI at 30 to 40 days and with phone survey at 6 months and 12 months.
  The secondary outcomes include the CMRI transmurality of scar, area at risk, myocardial salvage index, microvascular obstruction (MVO), left ventricle (LV) thrombus, and LV ejection fraction (EF). Important covariates include symptoms and ST segment resolution before and after the PCI, peak cardiac troponin (cTn), and angiographic TIMI flow and myocardial perfusion grade.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Study Director — WHC
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States